CLINICAL TRIAL: NCT00967213
Title: Changes in Preferential Hyperacuity Perimeter (PHP) and Fundus Autofluorescence (FAF) in Patients With Neovascular Age-related Macular Degeneration Receiving Combination of Ranibizumab and Verteporfin Therapy
Brief Title: Combination of Ranibizumab and Verteporfin Therapy in Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Korea Ltd. (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CBPD952AKR03; CCT-NAPN-18335
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

ARMS (1):
- Ranibizumab (Experimental): three session of monthly injection of Lucentis® (week 0, 4, 8). After 4 weeks from third injection, a session of verteporfin PDT (week 12) and fourth injection of Lucentis® (week 16) will be added at intervals of 4 weeks. Two more combined treatment with verteporfin PDT and Lucentis® injection 4 weeks apart can be added at the treating physician's discretion in 3-month intervals (week 28, week 40).
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — Lucentis® (ranibizumab) 0.3mg (0.05ml volume) intravitreal injection. Eligible patients will be initially received three session of monthly injection of Lucentis® (week 0, 4, 8). After 4 weeks from third injection, a session of verteporfin PDT (week 12) and fourth injection of Lucentis® (week 16) will be added at intervals of 4 weeks. Two more combined treatment with verteporfin PDT and Lucentis® injection 4 weeks apart can be added at the treating physician's discretion in 3-month intervals (week 28, week 40).
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to evaluate changes in preferential hyperacuity perimeter (PHP) and fundus autofluorescence (FAF) in patients with neovascular age-related macular degeneration receiving combination of ranibizumab (LucentisTM) and verteporfin (Visudyne®) therapy

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age ≥ 50 years old
* Patients with primary active subfoveal CNV secondary to AMD
* Baseline best-corrected visual acuity (BCVA) in the study eye was from 20/40 to 20/400 using ETDRS chart
* Characteristics of AMD lesion

  * predominantly or minimally classic, or occult
  * absence of prior subfoveal treatment for macular disease
  * total lesion size ≤ 9 optic disc areas, with CNV component ≥ 50% of the lesion (unless a serous pigment epithelial detachment was present, in which case < 50% CNV was acceptable)
  * active choroidal neovascularization leakage
  * submacular blood < 50% and subretinal fibrosis < 25% of the total lesion

Exclusion Criteria:

* additional eye disease that could compromise VA
* CNV unrelated to AMD
* ocular inflammation
* vitreous hemorrhage
* retinal hemorrhage (other than AMD related submacular blood) > 1 disc areas
* intraocular surgery ≤ 1 month before day 0
* uncontrolled glaucoma
* prior treatments with verteporfin PDT
* laser photocoagulation or other intervention for AMD
* previous treatment with external-beam radiation therapy or transpupillary thermotherapy
* history of vitrectomy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The change in ETDRS visual acuity letter scores from baseline. | every 4 weeks (up to 52 weeks)

SECONDARY OUTCOMES:
Effect on CNV and RPE using preferential hyperacuity perimeter (PHP) and fundus autofluorescence (FAF). Retinal thickness using optical coherence tomography (OCT). Recurrence of fluorescein leakage. The need for additional PDT treatment | every 4 weeks (up to 52 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Hyung-Woo Kwak, Principal Investigator — Dept. of ophthalmology, KyungHee Medical Center
Locations (1):
- Dept. of Ophthalmology, KyungHee Medical Center, #1 Hoegi, Dongdaemun-gu, Seoul, South Korea